CLINICAL TRIAL: NCT00197769
Title: Immunogenicity of a Reduced Primary Schedule for Pneumococcal Conjugate Vaccine in UK Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Public Health England (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PNC1/2
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2008-02

CONDITIONS: Streptococcus Pneumoniae

INTERVENTIONS:
Biological: 9 valent pneumococcal con jugate vaccine

SUMMARY:
The purpose of the trial is to determine the minimum of doses of a new nine valent pneumococcal conjugate vaccine required to protect UK infants and toddlers

DETAILED DESCRIPTION:
A new vaccine against pneumococcal infection is now available in the UK and has already been in routine use in the US for five years. The purpose of the trial is to determine the minimum number of does required to protect UK infants and toddlers, and to assess the compatibility of the pneumococcal vaccine with the other vaccines given in the UK childhood immunisation programme. The vaccine used in the US protects against seven strains of pnemococcus whereas the vaccine used in this trial protects against nine strains. Infants received either two doses at two and four months or three doses at two, three and four months of age, the latter comprising the routine infant schedule for other paediatric vaccines in the UK. The infants also received the usual vaccines against diphtheria , tetanus, polio, whooping cough and Hib together with meningitis C vaccine which is currently only used in the UK and a few other countries worldwide. A group of toddlers aged twelve to fifteen months also took apart and received either one or two doses of pneumococcal vaccine around the same time as their MMR vaccine. All children in the study received a booster dose some months later. The response to the vaccine is assessed by measuring levels of protective antibodies to the pneumococcal strains in blood samples taken at various times during the immunisation schedule.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by parent/guardian for receipt of study vaccines and for blood samples
* Age at first dose: Infants 7-11 weeks; toddlers 12-18 months

Exclusion Criteria:

* Previous bacteriologically confirmed pneumococcal or meningococcal disease
* Contraindications for pneumococcal, meningococcal, Hib, DTP, MMR immunisations as listed in the UK handbook, "Immunisation Against Infectious Disease" Edition 1996.
* Language difficulty in parents sufficient to preclude adequate comprehension of the information sheet, consent form and study nurses' explanation of the study
* Children participating in any other clinical trial
* Immunocompromised
* Acute systemic illness or fever > 38C on day of vaccination - deferral

Ages: 7 Weeks to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 2000-09; Study Completion 2004-01

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Miller, MBBS FRCPath, Principal Investigator — Public Health England

REFERENCES:
- [Result] Goldblatt D, Southern J, Ashton L, Richmond P, Burbidge P, Tasevska J, Crowley-Luke A, Andrews N, Morris R, Borrow R, Cartwright K, Miller E. Immunogenicity and boosting after a reduced number of doses of a pneumococcal conjugate vaccine in infants and toddlers. Pediatr Infect Dis J. 2006 Apr;25(4):312-9. doi: 10.1097/01.inf.0000207483.60267.e7. PMID 16567982